CLINICAL TRIAL: NCT00421642
Title: An Open-Label Study of the Human Anti-TNF Monoclonal Antibody Adalimumab in Ulcerative Colitis Patients
Brief Title: Open-Label Adalimumab for Ulcerative Colitis Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: William Sandborn, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-002167
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Adalimumab — The loading dose will be 160 mg. A dose of 80 mg will be given at Week 2 and 40 mg every other week starting at Week 4 until completion at Week 24. If it is found that they are not responding to 40 mg of adalimumab at Week 8 or later, the dose may be increased to 40 mg weekly.
  Other Names: Humira

SUMMARY:
This is an open-label study of 20 patients designed to demonstrate the safety, tolerability and preliminary evidence of benefit of adalimumab in the treatment of subjects with Ulcerative Colitis, both in patients who have never received anit-TNF agents and in those who have lost response or developed intolerance to previous infliximab therapy.

ELIGIBILITY:
Inclusion Criteria

1. Males and females 18 years of age and older
2. Female subjects must utilize a highly effective method of birth control throughout the study and for 70 days after study completion, or female subjects must not be of childbearing potential, defined as postmenopausal at least two years, or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
3. A diagnosis of UC for greater than 3 months.
4. UC diagnosis confirmed by endoscopy with exclusion of infectious cause.
5. Active ulcerative colitis with a Mayo Clinic Score (see Appendix C) of 6 to 12 points with moderately-to-severely active disease on sigmoidoscopy (endoscopic subscore of at least 2) despite concurrent treatment with corticosteroids, and/or azathioprine or 6 mercaptopurine and/or 5-aminosalicylate-containing medications. Patients who previously have not responded to or could not tolerate corticosteroids (within the past 18 months), or azathioprine or 6 mercaptopurine (both within the past 5 years), or 5 aminosalicylate-containing medications (within the past 18 months) will not required to be taking concurrent therapy at enrollment.
6. Either anti-TNF agent naïve or those with previous clinical response to infliximab therapy for UC with subsequent loss of response AND/OR are unable to tolerate further infliximab therapy for UC due to acute or delayed reactions, as defined by the investigator.
7. Subjects must be able and willing to give written informed consent and to comply with the requirements of this study protocol.
8. Adequate cardiac, renal and hepatic function as determined by principal investigator and demonstrated by screening laboratory evaluations, questionnaires, and physical examination results that are within normal limits.

Exclusion Criteria

1. History of cancer or lymphoproliferative disease other than a successfully and completely treated squamous cell or basal cell carcinoma of the skin.
2. Subjects with a history of Listeria, Hepatitis B infection, central nervous system (CNS) demyelinating disease, or human immunodeficiency virus (HIV) or a history of previously untreated TB. See Appendix B.
3. Subjects with Crohn?s Disease
4. Subjects with symptomatic obstructive strictures
5. Subjects who have had subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Kock pouch, or ileostomy for ulcerative colitis or are planning subtotal colectomy or colectomy within 8 weeks of starting the study medication.
6. Subjects who are currently receiving total parenteral nutrition (TPN).
7. Any investigational chemical agent in the past 30 days or 5 half-lives prior to screening (whichever is longer). Patients who have previously been treated with infliximab and responded, and then become intolerant to infliximab or lost response, can be treated >/= 4 weeks from their last infliximab dose.
8. Antibiotic treatment for any systemic infection within 3 weeks prior to screening.
9. Female subjects who are pregnant or breast-feeding.
10. History of clinically significant drug or alcohol abuse in the prior year.
11. Poorly controlled medical condition, including but not limited to diabetes with documented history of recurrent infections or cerebrovascular accidents (within 3 months).
12. Subjects who have been on cyclosporine or tacrolimus within 4 weeks of screening.
13. Subjects who have been on methotrexate within 4 weeks of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The Primary pilot efficacy variable will be the induction of clinical response, which is defined as a decrease in Mayo score less than 30% from baseline or less than 3 points PLUS decrease in rectal bleeding sub-score less than or equal to 1 at week 8 | 24 Weeks

SECONDARY OUTCOMES:
Clinical remission at each visit | 24 Weeks
Clinical response at each visit | 24 Weeks
Improvement in the mucosal inflammation at week 8 | 24 Weeks
Mayo Score | 24 Weeks
Ability to taper and discontinue steroids according to the tapering schedule after week 8 | 24 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: William J. Sandborn, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic, Scottsdale, Arizona
  - University of Chicago, Chicago, Illinois
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Result] Afif W, Leighton JA, Hanauer SB, Loftus EV Jr, Faubion WA, Pardi DS, Tremaine WJ, Kane SV, Bruining DH, Cohen RD, Rubin DT, Hanson KA, Sandborn WJ. Open-label study of adalimumab in patients with ulcerative colitis including those with prior loss of response or intolerance to infliximab. Inflamm Bowel Dis. 2009 Sep;15(9):1302-7. doi: 10.1002/ibd.20924. PMID 19408340